CLINICAL TRIAL: NCT00716170
Title: The Role of GIP, GLP-1 and GLP-2 in Type 2 Diabetic Hyperglucagonemia
Brief Title: GIP, GLP-1 and GLP-2 in Type 2 Diabetic Hyperglucagonemia
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Collaborators: University of Copenhagen (Other); The Danish Medical Research Council (Other); The Danish Diabetes Association (Other)
Responsible Party: Principal Investigator, Asger Lund, MD, Herlev Hospital
Other Study IDs: 1301831410
Record Dates: First submitted 2008-07-10; First posted 2008-07-16 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2009-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; Glucagon; Insulin; Incretin hormones; Glucose-dependent insulinotropic polypeptide; Glucagon-like peptide-1; Glucagon-like peptide-2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — Incretins; Glucagon-Like Peptide 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood plasma and leucocytes
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A:: Patients with type 2 diabetes mellitus
  Interventions: Biological: Glucose-dependent insulinotropic polypeptide (GIP), glucagon-like peptide-1 (GLP-1) and glucagon-like peptide-2 (GLP-2)

INTERVENTIONS:
Biological: Glucose-dependent insulinotropic polypeptide (GIP), glucagon-like peptide-1 (GLP-1) and glucagon-like peptide-2 (GLP-2) — Day A: Oral glucose tolerance test (50g glucose)
  Day B: Isoglycemic intravenous (iv) glucose infusion
  Day C: Isoglycemic iv glucose infusion + iv GIP infusion (0-20 min: 4 pmol/kg body weight/min; 20-50 min: 2 pmol/kg body weight/min)
  Day D: Isoglycemic iv glucose infusion + iv GLP-1 infusion (0-20 min: 0,6 pmol/kg body weight/min; 20-50 min: 0,3 pmol/kg body weight/min)
  Day E: Isoglycemic iv glucose infusion + iv GLP-2 infusion (0-20 min: 1 pmol/kg body weight/min; 20-50 min: 0,5 pmol/kg body wight/min)
  Day F: Isoglycemic iv glucose infusion + iv infusion of GIP, GLP-1 and GLP-2 in doses as Day C, D and E.
  Other Names: Human GIP (glucose-dependent insulinotropic polypeptide); Human GLP-1 (glucagon-like peptide-1); Human GLP-2 (glucagon-like peptide-2)

SUMMARY:
In order to investigate the mechanisms underlying the hyperglucagonemia characterizing patients with type 2 diabetes mellitus (T2DM) we wish to test the following hypothesis: Do pancreatic alpha-cells exhibit inappropriate glucagon responses to substances released from the small intestine (GIP, GLP-2 and GLP-2) in patients with T2DM?

DETAILED DESCRIPTION:
Patients with T2DM are not able to suppress their secretion of glucagon after a meal or after oral ingestion of glucose. Patients actually respond with pathological high plasmaglucagon concentrations to these stimuli. Previous studies have shown that postprandial hyperglucagonemia results in increased hepatic glucose production and therefore contributes significantly to the hyperglycemia characterizing these patients.

Recently we have shown that patients with T2DM exhibit a normal suppression of glucagon secretion following an adjustable intravenous (iv) glucose challenge mimicking the glucose excursion following a 50-g oral glucose tolerance test (OGTT) with the latter resulting in lack of glucagon suppression. Why this difference? A possible explanation could be that the oral administration stimulates intestinal factors resulting in a differentially glucagon response to the two similar glucose excursions. We wish to establish whether GIP, GLP-1 and/or GLP-2 are responsible for the inappropriate glucagon suppression following OGTT and meals in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians with diet and/or tablet treated T2DM of at least 3 months duration (diagnosed according to the criterias of the World Health Organization (WHO))
* Normal Hemoglobin
* Prior Informed Consent

Exclusion Criteria:

* Liver disease (ALAT/ASAT > 2 x upper normal value)
* Diabetic nephropathy (se-creatinin > 130 um and/or albuminuria
* Treatment with drugs that cannot be discontinued for 12 hours

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be recruted from the outpatient clinic of Department of Endocrinology, Herlev Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Plasma glucagon responses | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tina Vilsbøll, MD DMSc, Study Chair — Herlev Hospital; Filip K Knop, MD PhD, Study Director — Gentofte Hospital
Locations (1):
- Department of Endocrinology J, Herlev Hospital, Herlev, Herlev, Denmark

REFERENCES:
- [Background] Expert Committee on the Diagnosis and Classification of Diabetes Mellitus. Report of the expert committee on the diagnosis and classification of diabetes mellitus. Diabetes Care. 2003 Jan;26 Suppl 1:S5-20. doi: 10.2337/diacare.26.2007.s5. No abstract available. PMID 12502614
- [Background] Unger RH, Orci L. Glucagon and the A cell: physiology and pathophysiology (first two parts). N Engl J Med. 1981 Jun 18;304(25):1518-24. doi: 10.1056/NEJM198106183042504. No abstract available. PMID 7015132
- [Background] Unger RH, Orci L. Glucagon and the A cell: physiology and pathophysiology (second of two parts). N Engl J Med. 1981 Jun 25;304(26):1575-80. doi: 10.1056/NEJM198106253042604. No abstract available. PMID 7015135
- [Background] Shah P, Vella A, Basu A, Basu R, Schwenk WF, Rizza RA. Lack of suppression of glucagon contributes to postprandial hyperglycemia in subjects with type 2 diabetes mellitus. J Clin Endocrinol Metab. 2000 Nov;85(11):4053-9. doi: 10.1210/jcem.85.11.6993. PMID 11095432
- [Background] Knop FK, Vilsboll T, Madsbad S, Holst JJ, Krarup T. Inappropriate suppression of glucagon during OGTT but not during isoglycaemic i.v. glucose infusion contributes to the reduced incretin effect in type 2 diabetes mellitus. Diabetologia. 2007 Apr;50(4):797-805. doi: 10.1007/s00125-006-0566-z. Epub 2007 Jan 16. PMID 17225124
- [Background] Nauck MA, Homberger E, Siegel EG, Allen RC, Eaton RP, Ebert R, Creutzfeldt W. Incretin effects of increasing glucose loads in man calculated from venous insulin and C-peptide responses. J Clin Endocrinol Metab. 1986 Aug;63(2):492-8. doi: 10.1210/jcem-63-2-492. PMID 3522621
- [Background] Knop FK, Vilsboll T, Hojberg PV, Larsen S, Madsbad S, Volund A, Holst JJ, Krarup T. Reduced incretin effect in type 2 diabetes: cause or consequence of the diabetic state? Diabetes. 2007 Aug;56(8):1951-9. doi: 10.2337/db07-0100. Epub 2007 May 18. PMID 17513701
- [Background] Nauck MA, Kleine N, Orskov C, Holst JJ, Willms B, Creutzfeldt W. Normalization of fasting hyperglycaemia by exogenous glucagon-like peptide 1 (7-36 amide) in type 2 (non-insulin-dependent) diabetic patients. Diabetologia. 1993 Aug;36(8):741-4. doi: 10.1007/BF00401145. PMID 8405741
- [Background] Holst JJ. On the physiology of GIP and GLP-1. Horm Metab Res. 2004 Nov-Dec;36(11-12):747-54. doi: 10.1055/s-2004-826158. PMID 15655703
- [Background] Meier JJ, Gallwitz B, Siepmann N, Holst JJ, Deacon CF, Schmidt WE, Nauck MA. Gastric inhibitory polypeptide (GIP) dose-dependently stimulates glucagon secretion in healthy human subjects at euglycaemia. Diabetologia. 2003 Jun;46(6):798-801. doi: 10.1007/s00125-003-1103-y. Epub 2003 May 23. PMID 12764578
- [Background] Nauck MA, Heimesaat MM, Orskov C, Holst JJ, Ebert R, Creutzfeldt W. Preserved incretin activity of glucagon-like peptide 1 [7-36 amide] but not of synthetic human gastric inhibitory polypeptide in patients with type-2 diabetes mellitus. J Clin Invest. 1993 Jan;91(1):301-7. doi: 10.1172/JCI116186. PMID 8423228
- [Background] Vilsboll T, Krarup T, Madsbad S, Holst JJ. Defective amplification of the late phase insulin response to glucose by GIP in obese Type II diabetic patients. Diabetologia. 2002 Aug;45(8):1111-9. doi: 10.1007/s00125-002-0878-6. Epub 2002 Jul 4. PMID 12189441
- [Background] Meier JJ, Nauck MA, Pott A, Heinze K, Goetze O, Bulut K, Schmidt WE, Gallwitz B, Holst JJ. Glucagon-like peptide 2 stimulates glucagon secretion, enhances lipid absorption, and inhibits gastric acid secretion in humans. Gastroenterology. 2006 Jan;130(1):44-54. doi: 10.1053/j.gastro.2005.10.004. PMID 16401467
- [Background] Schmidt WE, Siegel EG, Creutzfeldt W. Glucagon-like peptide-1 but not glucagon-like peptide-2 stimulates insulin release from isolated rat pancreatic islets. Diabetologia. 1985 Sep;28(9):704-7. doi: 10.1007/BF00291980. PMID 3905480
- [Background] Sorensen LB, Flint A, Raben A, Hartmann B, Holst JJ, Astrup A. No effect of physiological concentrations of glucagon-like peptide-2 on appetite and energy intake in normal weight subjects. Int J Obes Relat Metab Disord. 2003 Apr;27(4):450-6. doi: 10.1038/sj.ijo.0802247. PMID 12664078